CLINICAL TRIAL: NCT07385404
Title: Factors Contributing to Readmission of Heart Failure Patients to Emergency Departments and Prospects for Improvement
Acronym: CARDIO-REA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-04-Obs-CHRMT
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Readmissions
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) represents a major public health challenge due to its increasing prevalence and significant impact on healthcare systems.

The burden of frequent readmissions leads to increased healthcare costs, deterioration in the quality of care, and reduced availability of hospital resources for new patients. It is therefore essential to optimize the management of patients with heart failure from their first visit to the emergency department in order to improve their prognosis and reduce the risk of rehospitalization.

In this context, this study aims to identify the key factors associated with early readmissions (< 30 days) and to propose strategies to improve patient management and follow-up after discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, admitted to the emergency department for confirmed acute heart failure. Hospitalization following admission to the emergency department, with at least one documented post-hospitalization follow-up visit.

Exclusion Criteria:

* Patients under the age of 18 with a primary diagnosis unrelated to heart failure after analysis of their medical records. Patients in palliative care receiving only comfort treatment. No documented post-hospitalization follow-up. Patients who object to the use of their medical data for research purposes.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized for acute heart failure over a period of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Key factors determining the rehospitalization | 6 months
  Key factors determining the rehospitalization of patients with heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Laure ABENSUR VUILLAUME, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No